CLINICAL TRIAL: NCT04288453
Title: The Impact of Participation on Body Functions Among Youth With Physical Disabilities: A Pragmatic Individual-based Study
Brief Title: The Impact of Participation on Body Functions Among Youth With Physical Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other); Drexel University (Other)
Responsible Party: Principal Investigator, Dana Anaby, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 419713
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy; Spina Bifida; Musculoskeletal Disorders
Keywords: participation; environmental barriers; youth; disabilities; body functions
MeSH Terms: conditions — Cerebral Palsy; Spinal Dysraphism; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: A 22-week interrupted time series design with multiple baselines systematically replicated across 30 youth with physical disabilities will be employed.
Masking Description: Assessors will be blinded to the time point in which the intervention begins and to the chosen activity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based activity program (Experimental): Engagement in 8-week community-based activity program
  Interventions: Behavioral: Engagement in a 8-week community-based activity program

INTERVENTIONS:
Behavioral: Engagement in a 8-week community-based activity program — Participants engage in a 8-week community-based activity program of their choice. In order to engage in the selected activity, an Occupational Therapist (OT) will meet with each youth in their home. Using the PREP 5 steps (Make goals; Map out a plan; Make it happen; Measure the process and outcomes; Move forward) the youth will choose a community program. The OT will then search for the appropriate program, identify and remove potential environmental barriers for participation in that activity (e.g., accessibility, equipment) and educate program instructors regarding the youth's specific needs. This process, which includes up to 12 hours of working with the OT, will set the stage for enrolment of the youth in a community program for a period of 8 weeks - the actual intervention phase.
  Other Names:
  • Pathways and Resources for Engagement and Participation

SUMMARY:
Youth with physical disabilities experience greater limitations to participation in community- based activities than do their average-developing peers, which can result in poor health outcomes. Emerging treatment approaches aimed at improving activity and participation have shifted from focusing only on impaired body functions towards the performance of functionally meaningful activities within the youth's natural environment. It is unclear; however, whether targeting intervention at the activity/participation level can simultaneously result in improvement of personal functional skills (e.g., reaching) and body functions (e.g., range of motion, balance) - components known to worsen with age and, thus, important to address and maintain within the rehabilitation process. Our team has partnered with key community-based stakeholders including youth, clinicians and policy-makers, and together we plan to examine whether engaging in an 8-week self-chosen community-based activity (e.g., sledge hockey, boccia) can lead to a significant improvement in three key body functions: motor, cognitive and affective. Thirty youth with physical disabilities will take part in the study and engage in an activity program of their choice. Changes in their body functions (e.g., movement, attention, mood) will be measured multiple times before, during and after engagement in the chosen activity/program. Findings of this study can guide clinicians, families and policy-makers to select effective approaches that not only promote participation but also facilitate additional motor and mental benefits from one single intervention. Such treatment approaches may also reduce the burden on the healthcare system as well as on the youth and families. Moreover, findings can advance our understanding of methods for testing complex and unique 'real-life' individual-based interventions that are highly relevant to practice.

DETAILED DESCRIPTION:
Youth with physical disabilities experience restrictions to participation in community-based activities, leading to poor health outcomes. Personalized participation-based treatment approaches, implemented in the individual's natural environment, are considered recommended practice. However, it is unclear whether enhancing participation (e.g., engaging in sledge hockey) can simultaneously improve both body functions (e.g., grip, trunk control) and activity performance - two key outcomes in pediatric rehabilitation. Specifically, the impact of participation in a self-chosen real-life activity, that is meaningful to the youth, on a range of functions (motor, cognitive and affective) has not been established. Supported by Canadian Institutes of Health Research (CIHR), we first proved the effectiveness of the Pathways and Resources for Engagement and Participation (PREP) intervention in promoting youth's community participation; then, through Strategy for Patient-Oriented Research (SPOR), we successfully pilot- tested an innovative pragmatic clinical trial to improve body functions through participation, informing the design of this proposed larger study. Using the PREP, we aim to examine the impact of youth engagement in an 8-week community-based activity program (e.g., drawing, swimming) on underlying body functions or impairments (e.g., movement, attention, mood), as well as on performance of the selected activity. Specifically, change in 3 relevant body functions will be examined: motor (using the Functional Reach Test, Trunk Impairment Scale, and dynamometer), cognitive and affective (using the Behavior Assessment System for Children), and activity performance (via the Canadian Occupational Performance Measure). A 22-week interrupted time series design with multiple baselines systematically replicated across 30 youth with physical disabilities (e.g., cerebral palsy, spina bifida) aged 15 to 24 will be employed. Each activity, individually selected by the youth, will be analyzed using the task analysis approach to identify underlying body functions. These functions will be measured multiple times throughout the entire study, resulting in 90 trajectories of change in body functions (30 youth X 3 functions) and 30 trajectories representing change in activity performance. A linear model will be fit for each of the 120 trajectories. Motor-related scores will be standardized to allow comparison across different outcomes and mixed-effects models will be used to estimate an intervention effect across participants. Our interdisciplinary team includes researchers in the field of childhood disability, including occupational therapy, physical therapy and pediatric medicine. Partnered with the Centre of Integrated University Health and Social Services (CIUSSS) West-Central Montreal and CanChild Centre for Childhood Disability, as well as key local and national stakeholders, the team will collaborate throughout the research process. This novel patient-oriented study will support a paradigm shift in clinical practice and build knowledge that can guide clinicians, families and policy-makers in appraising the benefits of participation- based therapies on improving both functional capacities and performance in meaningful life activities. Describing the multiple benefits generated by one single intervention can facilitate efficient youth-engaging therapies, contributing to the provision of pediatric rehabilitation services. Findings can also enhance knowledge of pragmatic clinical trials for testing complex individual-based interventions highly applicable to practice.

ELIGIBILITY:
Inclusion Criteria:

* have a physical disability (e.g., cerebral palsy, spina bifida, musculoskeletal disorders)
* restricted mobility, such as an inability to navigate all surfaces and stairs independently and safely without the use of aids, physical assistance or external support

Exclusion Criteria:

Youth who are recovering within the first year following a severe brain injury or an orthopedic surgery or botulinum toxin treatment 6 months prior or anticipated during the study period or those with degenerative disorders will be excluded.

Youth with significant intellectual delay will be excluded due to the demands required for completing self-reported assessments.

Youth with co-occurrence of an untreated mental health condition will also be excluded.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Behavioral Assessment System for Children | 22 weeks
  Evaluates cognitive and affective body functions using a 4-point scale. T-scores range from 0 to 120 in which lower scores indicate greater cognitive and affective body functions.
Trunk Impairment Scale | 22 weeks
  Assesses trunk control and includes 3 sub-scales; static sitting balance, dynamic sitting balance and coordination. It contains 17 items rated on a 2-, 3- or 4- point scale. Total score measures motor body functions in terms of trunk control. Total score ranges from 0 (low performance) to 23 (high performance).
Functional Reach Test | 22 weeks
  Assesses motor body functions in terms of reaching. The maximum distance in inches the participant can reach forward while standing/sitting in a fixed position is measured; units: inches.
Jamar/Handheld micro Force Evaluation and Testing 2 (microFET2) Dynamometers | 22 weeks
  Measures motor body functions in terms of maximal grip, pinch strength and isometric muscle strength; units: pounds of force. Scores range from 0 to 200 pounds.
Goniometer | 22 weeks
  Measures active range of motion of specific joints relevant to the activity and based on the task analysis; units: degrees of range of motion.
Canadian Occupational Performance Measure | 22 weeks
  10-point scale that measures activity performance. Score ranges from 1 (unable to perform) to 10 (performs extremely well).

OTHER OUTCOMES:
Life-Habits (LIFE-H) | This outcome will be assessed once at baseline only (week 1).
  Evaluates participation accomplishments in daily activities and social roles using a 4-point scale. Scores range from 1 (not accomplished) to 4 (accomplished with no difficulty).

CONTACTS AND LOCATIONS:
Overall Officials: Dana Anaby, PhD, Principal Investigator — McGill University
Locations (1):
- Lethbridge-Layton-Mackay Rehabilitation Center of CIUSSS West-Central Montreal (Mackay site), Montreal, Quebec, Canada